CLINICAL TRIAL: NCT06881342
Title: Evaluating the Feasibility of a School-based Stepped Care Program for Internalizing Symptoms in Adolescents in Pakistan
Acronym: SMART-STEP
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Global Institute of Human Development (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Treatment
Other Study IDs: GIHD/Trials/2024/01; R01MH131025-03 (NIH)
Record Dates: First submitted 2025-03-05; First posted 2025-03-18 (Actual); Last update posted 2025-04-22 (Actual); Status verified 2025-04

CONDITIONS: Depression, Anxiety; Distress, Emotional; Psychosocial Problem; Functioning, Psychosocial
MeSH Terms: conditions — Depression; Anxiety Disorders

STUDY DESIGN:
Intervention Model Description: In this pilot sequential multiple assignment cluster randomized controlled trial, randomization will occur in two stages. First, school clusters (N=8), stratified by sex, will be randomized to intervention or control arms in a 1:1 allocation ratio. Schools in the intervention arm will receive the Enhanced School Mental Health Program (eSMHP) Plus by teachers and non-specialists in classroom settings. It aims at improving providers' mental health literacy, enabling early identification and management of socioemotional issues in adolescents, and enhancing teachers' well-being. Adolescents in the control arm will receive Enhanced Treatment as Usual (ETAU), which is eSMHP delivered by teachers only. At 6 weeks from baseline, a second randomization will occur at the individual level based on gender and PSC scores. In both arms, adolescents scoring ≥28 on PSC will be re-randomised to continue initial treatment (eSMHP Plus or eSMHP) or a step-up CBT-based guided self-help app.
Who Masked: Investigator, Outcomes Assessor
Masking Description: Participants will not be blinded to treatment allocation. However, all outcome measures will be administered by researchers' blind to allocation status. It is not possible to blind adolescents, caregivers, intervention facilitators, intervention supervisors, data managers, or the trial manager to the treatment allocation because of the nature of the intervention. The assessors, trial statistician, and investigator(s) will be blind to treatment allocation status. To ensure masking during the trial, the intervention and assessment teams will be based at separate office locations and will not have any interaction. The assessment team members will also be non-residents of the study place. Furthermore, participants will be each individually instructed not to disclose their treatment allocation status to the assessors during any follow-up assessments. The fidelity of masking will be measured by having assessors guess the condition of each participant at the end of each assessment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention arm - Enhanced School Mental Health Program (eSMHP) Plus (Experimental): The first-stage intervention, eSMHP Plus, is delivered by teachers and non-specialists in classrooms. eSMHP enhances mental health literacy, training providers in early identification, counseling, life skills, positive discipline, parental engagement, referrals, and teacher well-being. Teachers follow a lesson plan, supported by non-specialists through biweekly school visits. Non-specialists co-deliver activities and supervise teachers to address challenges and promote well-being. At six weeks, adolescents scoring ≥28 on PSC are re-randomized to continue eSMHP Plus or receive a step-up, CBT-based guided self-help app for two months. The app, accessible via tablet/mobile, is based on empirically supported strategies.
  Interventions: Behavioral: Enhanced School Mental Health Program (eSMHP)
- Enhanced Treatment-as-usual (Active Comparator): The first-stage intervention in the control arm, eSMHP, is delivered by teachers only. Teachers in ETAU complete online training (www.learnwithshine.org) to enhance mental health literacy, learning to identify socioemotional issues and provide basic psychosocial support through counseling skills, life skills, positive discipline, parental engagement, and referrals. A dedicated module promotes teacher well-being. At six weeks, adolescents scoring ≥28 on PSC are re-randomized to continue eSMHP or receive a step-up, CBT-based guided self-help app for two months. The app, accessible via tablet/mobile, is based on empirically supported strategies and offers comprehensive features for adolescents.
  Interventions: Behavioral: Enhanced School Mental Health Program (eSMHP)

INTERVENTIONS:
Behavioral: Enhanced School Mental Health Program (eSMHP) — The first-stage intervention is eSMHP Plus in the intervention arm and eSMHP in the control arm. In the intervention arm, adolescents receive eSMHP Plus from teachers and non-specialists, while in the control arm, they receive eSMHP from teachers. eSMHP, based on developmental, behavioral, social, and cognitive theories, enhances teachers' mental health literacy, training them in early identification, basic counseling, life skills, positive discipline, parental engagement, referrals, and teacher well-being. The second-stage intervention is a CBT-based self-help app. At six weeks, adolescents scoring ≥28 on PSC in both arms (indicating psychosocial distress) are re-randomized to continue their initial treatment (eSMHP Plus or eSMHP) or receive a step-up, CBT-based guided self-help app for two months.
  Other Names: CBT-based Guided Self-Help Application

SUMMARY:
This study aims to explore effective ways to reduce depressive symptoms in adolescents through two school-based interventions. This study examines whether the Enhanced School Mental Health Program (eSMHP) Plus, delivered by teachers and non-specialists, can serve as a first-line intervention to reduce psychosocial distress-an intermediate outcome that must be addressed to lower the risk of depression (primary outcome) in adolescents. For those who do not respond to eSMHP Plus, the study investigates if a Cognitive Behavioural Therapy (CBT) based guided self-help app could be an effective step-up or second-level intervention. Researchers will assess the feasibility and acceptability of these approaches among 200 adolescents (aged 13-15) from 8 public schools in Rawalpindi, Pakistan. Findings will guide future large-scale studies and strategies for personalised mental health care for adolescents in low-resource settings.

DETAILED DESCRIPTION:
Background:

Internalizing symptoms among adolescents can have long-term devastating impacts on their lives unless they are identified and treated early and effectively. Both universal and indicated school-based interventions are recommended to address internalizing symptoms among adolescents. However, determining the optimal timing and dosage of these interventions remains a crucial question for effective adolescent mental healthcare. The investigators will conduct a pilot Sequential Multiple Assignment Randomized Controlled Trial (SMART) to explore the feasibility and acceptability of two evidence-informed intervention strategies (universal and indicated interventions) within the stepped care model, compare their timing and dosage, and determine in which sequence these interventions should be delivered to whom. This study aims to answer the question, "What works, for whom, under what conditions, and why, for internalizing symptoms in adolescents with a focus on depressive symptoms?"

Methods:

A 20-week single-blind pilot cluster SMART study will be conducted in 8 public schools in Rawalpindi, Pakistan, to assess the feasibility and acceptability of 2 intervention strategies (i.e., 1. teachers plus non-specialist delivered universal intervention called Enhanced School Mental Health Program [eSMHP] Plus and 2. Guided self-help application of Cognitive Behavioural Therapy-based indicated intervention to reduce depression (internalising symptoms) in adolescents. The study participants will be approximately 200 adolescents, aged 13-15 of both sexes, with psychosocial distress. Data on the feasibility and acceptability of the study design, views about augmented intervention options and procedures, and treatment response rates will be collected. Results from the pilot study will yield additional research questions and will improve our ability to successfully conduct the definitive SMART to inform personalised interventions for internalising symptoms in adolescents.

Discussion: The findings of the study will be used to inform the design of a subsequent fully powered, definitive SMART study in Pakistan.

ELIGIBILITY:
Inclusion Criteria:

1. Adolescents aged 13-15 years, studying in grades 7 and 8 of participating schools, provide assent and parental consent for participation in the study and screen positive for psychosocial distress on youth reported PSC (total score ≥ 28).

Exclusion Criteria:

1. Adolescents who require immediate in-patient (medical and/or psychiatric) care
2. Adolescents with acute protection risks as assessed by a researcher applying the definitions in the WHO mhGAP intervention guide.

Ages: 13 Years to 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 137 (Actual)
Dates: Start 2025-03-28 (Actual); Primary Completion 2025-06-30 (Estimated); Study Completion 2025-08-31 (Estimated)

PRIMARY OUTCOMES:
Patient Health Questionnaire (PHQ-9) for adolescents | Enrollment, and 6 weeks and 3-months from baseline
  Patient Health Questionnaire (PHQ-9) for adolescents is a 9-item instrument (on a 4-point Likert scale; range 0-27) to measure depressive symptoms in the past 2 weeks (Richardson et al., 2010) and that is previously adapted, validated and shown high reliability in Pakistan (Cronbach α=0.83).

SECONDARY OUTCOMES:
Pediatric Symptoms Checklist (PSC) | Enrollment, and 6 weeks and 3-months from baseline
  PSC will also serve as an intermediate tailoring variable. It is well-established 35-item scale. It consists of three subscales, internalizing, externalizing and attention problems. The Urdu version has been previously adapted and used in Pakistan, showing satisfactory reliability and validity.
Revised Children's Anxiety and Depression Scale (RCADS) | From enrollment to the end of treatment at 3-months
  It is a 25-item instrument (on a 4-point Likert scale; range 0-100) to measure levels of anxiety and low mood. It has two subscales (anxiety & depression). It has been adapted and used successfully in Pakistan.
Diagnostic and Statistical Manual of Mental Disorders (DSM)-5 Level 1 Cross-Cutting Symptom Measure | From enrollment to the end of treatment at 3-months
  It is a self-rated measure that assesses mental health domains that are important across psychiatric diagnoses. It is intended to help identify additional areas of inquiry that may have a significant impact on the child's treatment and prognosis. Each item on the measure is rated on a 5-point scale (0=none or not at all; 1=slight or rare, less than a day or two; 2=mild or several days; 3=moderate or more than half the days; and 4=severe or nearly every day). A rating of mild (i.e., 2) or greater on any item within a domain (except for suicidal ideation and psychosis) will serve as a guide for additional inquiry and follow-up to determine if a more detailed assessment for that domain is necessary.
Checklist of Somatic Symptoms of Distress | From enrollment to the end of treatment at 3-months
  It is a 10-item tool (on a 3-point Likert scale); 0-20 to measure somatic symptoms of distress. It has been previously adapted and used in Pakistan.
Experience of bullying | From enrollment to the end of treatment at 3-months
  Experience of bullying in the past 30 days will be measured through the contextualised version of the Bullying Victimization Questionnaire. The total score can range from 0 to 12, with higher scores indicating higher levels of victimization by peers.
School climate | From enrollment to the end of treatment at 3-months
  The change in school climate (students' relationship with teachers, belongingness with the schools and peers, students' commitment to the school tasks, and participation in school activities) will be measured using the adapted version of the Beyound Blue School Climate Questionnaire. The tool will be administered to both children and their caregivers. The questionnaire consists of 28 items. Each item is rated on a 3-point Likert scale (yes=1, No = 0, I can't say = no score). The total score of BBSCQ can range from 0 to 28, where higher scores indicate a more favourable view of the school climate.
Annual academic performance and classroom attendance questionnaire | From enrollment to the end of treatment at 3-months
  A study-specific questionnaire will be developed to obtain records of attendance and academic grades from the school records at baseline and 3 months post-intervention delivery.
Wellbeing | From enrollment to the end of treatment at 3-months
  Short Warwick Edinburgh Mental Wellbeing Scale (SWEMWS): It is a 7-item scale and assesses the mental wellbeing by evaluating the functioning of thoughts and feelings in the past two weeks. Items are rated on Likert scale that ranges from "none of the time" to "all of the time". The total score is calculated by summing the responses on all the items.
Teachers' wellness | From enrollment to the end of treatment at 3-months
  The Self Reporting Questionnaire (SRQ) is a 20-item self-report measure to detect non-specific psychological distress, developed by the WHO. Psychological distress is represented by subscales of physical symptoms and emotional symptoms. The SRQ items are scored 0 or 1. A score of 1 indicates the presence of symptoms of psychological distress
Teachers' sense of self-efficacy | From enrollment to the end of treatment at 3-months
  The 12 items Teachers Sense of efficacy scale will be used to assess teacher's belief about his or her capabilities to enhance students' learning and to be able to support students who are difficult or unmotivated. The scale measures teacher's efficacy on three subscales namely, instructional strategies, student engagement, and classroom management. The items are rated on 5 points Likert scale ranging from (1) 'None at all' to (5) 'A great deal'.
Psychosocial Profile of the School | From enrollment to the end of treatment at 3-months
  Each question is scored on a scale from 1 to 4, with 1 representing the lowest and 4 the highest rating of social and emotional support. To obtain an overall mean or average, the scores of all the answered questions are added and divided by the total number of questions answered. Higher scores indicate a better psychosocial environment at the school.
Caregivers' Wellbeing | From enrollment to the end of treatment at 3-months
  The Self Reporting Questionnaire (SRQ) is a 20-item self-report measure to detect non-specific psychological distress, developed by the WHO. Psychological distress is represented by subscales of physical symptoms and emotional symptoms. The SRQ items are scored 0 or 1. A score of 1 indicates the presence of symptoms of psychological distress
Alabama Parenting Questionnaire (APQ) | From enrollment to the end of treatment at 3-months
  The positive involvement subscale of the Alamaba Parenting Questionnaire (APQ) will be used to measure parenting practices. The subscale measures whether parents talk more friendly with children; help children in planning and conducting special activities; know what they are doing in their free time; play games with them; help them with their homework; get interested in their day-to-day plans and activities; and know about their friends. Items are rated on a five-point Likert scale (1 = never to 5 = almost always). The total score is calculated by summing all the items. The minimum score is 10, and the maximum score is 50. Higher scores indicate more positive outcomes.

CONTACTS AND LOCATIONS:
Overall Officials: Syed Usman Hamdani, PhD MBBS, Principal Investigator — Global Institute of Human Development
Locations (1):
- Global Institute of Human Development, Rawalpindi, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: Undecided
The availability of individual participant data (IPD) has not been determined at this time.

REFERENCES:
- [Background] Lei H, Nahum-Shani I, Lynch K, Oslin D, Murphy SA. A "SMART" design for building individualized treatment sequences. Annu Rev Clin Psychol. 2012;8:21-48. doi: 10.1146/annurev-clinpsy-032511-143152. Epub 2011 Dec 12. PMID 22224838
- [Background] Hamdani, S. U., Muzaffar, N., Huma, Z.E, Hamdani, A., Rauf, R., Farzeen, M., ... & Rahman, A. (2019). Using technology to advance school mental health: Experience from the Eastern Mediterranean Region Journal of the American Academy of Child & Adolescent Psychiatry, 58(10), S22.
- [Background] Hamdani SU, Huma ZE, Tamizuddin-Nizami A, Baneen UU, Suleman N, Javed H, Malik A, Wang D, Mazhar S, Khan SA, Minhas FA, Rahman A. Feasibility and acceptability of a multicomponent, group psychological intervention for adolescents with psychosocial distress in public schools of Pakistan: a feasibility cluster randomized controlled trial (cRCT). Child Adolesc Psychiatry Ment Health. 2022 Jun 21;16(1):47. doi: 10.1186/s13034-022-00480-z. PMID 35729589
- [Background] Hamdani SU, Huma ZE, Malik A, Tamizuddin-Nizami A, Javed H, Minhas FA, Jordans MJD, Sijbrandij M, Suleman N, Baneen UU, Bryant RA, van Ommeren M, Rahman A, Wang D. Effectiveness of a group psychological intervention to reduce psychosocial distress in adolescents in Pakistan: a single-blind, cluster randomised controlled trial. Lancet Child Adolesc Health. 2024 Aug;8(8):559-570. doi: 10.1016/S2352-4642(24)00101-9. PMID 39025557
- [Background] Hamdani, S., Huma, Z.E., Javed, H., Warraitch, A., Rahman, A., Nizami, A., & Minhas, F. (2021). Prevalence of psychosocial distress in school going adolescents in rural Pakistan: Findings from a cross-sectional epidemiological survey. BJPsych Open, 7(S1), S56-S57. doi:10.1192/bjo.2021.196
- [Background] Naveed S, Waqas A, Memon AR, Jabeen M, Sheikh MH. Cross-cultural validation of the Urdu translation of the Patient Health Questionnaire for Adolescents among children and adolescents at a Pakistani school. Public Health. 2019 Mar;168:59-66. doi: 10.1016/j.puhe.2018.11.022. Epub 2019 Jan 25. PMID 30685600
- [Background] Spence SH. Structure of anxiety symptoms among children: a confirmatory factor-analytic study. J Abnorm Psychol. 1997 May;106(2):280-97. doi: 10.1037//0021-843x.106.2.280. PMID 9131848
- [Background] Hamdani SU; Zill-e-Huma; Warraitch A, Suleman N, Muzzafar N, Minhas FA; F.R.C.Psych; Nizami AT; F.C.P.S.; Sikander S; F.C.P.S.; Pringle B, Hamoda HM, Wang D, Rahman A, Wissow LS. Technology-Assisted Teachers' Training to Promote Socioemotional Well-Being of Children in Public Schools in Rural Pakistan. Psychiatr Serv. 2021 Jan 1;72(1):69-76. doi: 10.1176/appi.ps.202000005. Epub 2020 Aug 25. PMID 32838678
- [Background] Shaffer D, Gould MS, Brasic J, Ambrosini P, Fisher P, Bird H, Aluwahlia S. A children's global assessment scale (CGAS). Arch Gen Psychiatry. 1983 Nov;40(11):1228-31. doi: 10.1001/archpsyc.1983.01790100074010. PMID 6639293
- [Background] Hamdani SU, Huma ZE, Wissow L, Rahman A, Gladstone M. Measuring functional disability in children with developmental disorders in low-resource settings: validation of Developmental Disorders-Children Disability Assessment Schedule (DD-CDAS) in rural Pakistan. Glob Ment Health (Camb). 2020 Jul 13;7:e17. doi: 10.1017/gmh.2020.10. eCollection 2020. PMID 32913656
- [Background] D'Zurilla, T. J., Nezu, A. M., & Maydeu-Olivares, A. (1999). Manualfor the Social Problem-Solving Inventory-Revised. North Towanda, NY: Multi-Health Systems
- [Background] Clarke DE, Kuhl EA. DSM-5 cross-cutting symptom measures: a step towards the future of psychiatric care? World Psychiatry. 2014 Oct;13(3):314-6. doi: 10.1002/wps.20154. No abstract available. PMID 25273306
- [Background] Jellinek MS, Murphy JM, Robinson J, Feins A, Lamb S, Fenton T. Pediatric Symptom Checklist: screening school-age children for psychosocial dysfunction. J Pediatr. 1988 Feb;112(2):201-9. doi: 10.1016/s0022-3476(88)80056-8. PMID 3339501
- [Background] Richardson LP, McCauley E, Grossman DC, McCarty CA, Richards J, Russo JE, Rockhill C, Katon W. Evaluation of the Patient Health Questionnaire-9 Item for detecting major depression among adolescents. Pediatrics. 2010 Dec;126(6):1117-23. doi: 10.1542/peds.2010-0852. Epub 2010 Nov 1. PMID 21041282
- [Background] Varni JW, Seid M, Rode CA. The PedsQL: measurement model for the pediatric quality of life inventory. Med Care. 1999 Feb;37(2):126-39. doi: 10.1097/00005650-199902000-00003. PMID 10024117
- See also: PedsQLTM. (2021). Measurement Model for the Pediatric Quality of Life Inventory. — http://www.pedsql.org/about_pedsql.html